CLINICAL TRIAL: NCT02658721
Title: Effects of Addition of Systemic Tramadol or Adjunct Tramadol to Lidocaine Used for Intravenous Regional Anesthesia in Patients Undergoing Hand Surgery
Brief Title: Effects of Systemic or Adjunct Tramadol Addition to Lidocaine Used for IVRA in Patients Undergoing Hand Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Abdulkadir Yektas, Dr. Abdulkadir Yektas, Bagcilar Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IVRA
Record Dates: First submitted 2015-12-10; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Anesthesia
Keywords: Systemic Tramadol; Adjunct Tramadol; Lidocain
MeSH Terms: interventions — Lidocaine; Tramadol; Fentanyl; Atropine; Midazolam; Diclofenac; Ephedrine; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- lidocaine+adjunct tramadol (Experimental): In the first group (LDC+TRA group), IVRA was performed with 3 mg/kg lidocaine (10% Lidocaine) plus 50 mg tramadol, which were administered after diluting with saline to 40 mL. While performing IVRA, 30 mL saline was simultaneously administered to the systemic circulation.
  Interventions: Drug: lidocaine+adjunct tramadol; Drug: Fentanyl; Drug: Atropine; Drug: Midazolam; Drug: Diclofenac sodium; Drug: Ephedrine; Drug: Ondansetron
- lidocaine+systemic tramadol (Experimental): In the second group (LDC+SysTRA group), IVRA was performed with 3 mg/kg lidocaine, which was diluted with saline to 40 mL. While performing IVRA, 50 mg tramadol diluted with saline to 30 mL was simultaneously administered to the systemic circulation.
  Interventions: Drug: lidocaine+systemic tramadol; Drug: Fentanyl; Drug: Atropine; Drug: Midazolam; Drug: Diclofenac sodium; Drug: Ephedrine; Drug: Ondansetron
- lidocaine (Active Comparator): In the third group (LDC group), IVRA was performed with 3 mg/kg lidocaine, which was diluted with saline to 40 mL.
  Interventions: Drug: Lidocaine; Drug: Fentanyl; Drug: Atropine; Drug: Midazolam; Drug: Diclofenac sodium; Drug: Ephedrine; Drug: Ondansetron

INTERVENTIONS:
Drug: Lidocaine
  Arms: lidocaine
Drug: lidocaine+adjunct tramadol — IVRA was performed with 3 mg/kg lidocaine (10% Lidocaine) plus 50 mg tramadol, which were administered after diluting with saline to 40 mL. While performing IVRA, 30 mL saline was simultaneously administered to the systemic circulation
  Other Names: tramadol
  Arms: lidocaine+adjunct tramadol
Drug: lidocaine+systemic tramadol — IVRA was performed with 3 mg/kg lidocaine, which was diluted with saline to 40 mL. While performing IVRA, 50 mg tramadol diluted with saline to 30 mL was simultaneously administered to the systemic circulation
  Other Names: tramadol
  Arms: lidocaine+systemic tramadol
Drug: Fentanyl — If the patient had a VAS score of >4 and if required, 1 μg/kg fentanyl was administered for analgesia and the dosage and time were recorded.
Drug: Atropine — The patients received premedication 45 min before the surgery with intramuscular 0.01 mg/kg atropine.
  In case of bradycardia (HR <50/min), 0.5 mg intravenous atropine was administered.
Drug: Midazolam — The patients received premedication 45 min before the surgery with intramuscular 0.07 mg/kg midazolam
Drug: Diclofenac sodium — The patients with a VAS score of >4 were administered with 75 mg diclofenac sodium via intramuscular route.
Drug: Ephedrine — In the event of hypotension (systolic arterial pressure <90 mmHg or a decrease of more than 50 mmHg from the normal value) during the surgery, 5 mg intravenous ephedrine was administered.
Drug: Ondansetron — Intravenous 4 mg ondansetron was administered for nausea and vomiting.

SUMMARY:
Intravenous regional anesthesia (IVRA) is used in outpatient hand surgery as an easily applicable and cost-effective technique with clinical advantages. Nevertheless, IVRA has some disadvantages including anesthetic toxicity, slow-onset, poor muscle relaxation, tourniquet pain, and minimal postoperative pain relief. Providing an ideal anesthesia by overcoming these disadvantages is possible with the addition of some adjunct agents into local anesthetic substances. One of these adjunct agents used for IVRA is tramadol, a synthetic analgesic having opioid and nonopioid characteristics. The present study aimed to investigate the effects of addition of systemic tramadol or adjunct tramadol to lidocaine for IVRA in patients undergoing hand surgery..

DETAILED DESCRIPTION:
The present study included American Society of Anesthesiologists (ASA) I-II patients (n=60) who were planned to undergo hand surgery. Patients with Raynaud's disease, those with sickle-cell anemia, and those receiving any drug for history of allergy were excluded. Approval of the ethics committee and informed consents of the patients were obtained for the study.

According to a computer-generated randomization list, the patients were divided into three groups, containing 20 subjects in each. In the first group, Lidocaine (LDC)+Adjunct Tramadol (TRA), IVRA was performed with 3 mg/kg lidocaine (10% Lidocaine) plus 50 mg tramadol, which were administered after diluting with saline to 40 mL. While performing IVRA, 30 mL saline was simultaneously administered to the systemic circulation. In the second group, lidocaine (LDC)+systemic tramadol (SysTRA), IVRA was performed with 3 mg/kg lidocaine, which was diluted with saline to 40 mL. While performing IVRA, 50 mg tramadol diluted with saline to 30 mL was simultaneously administered to the systemic circulation. In the third group (LDC group), IVRA was performed with 3 mg/kg lidocaine, which was diluted with saline to 40 mL. While performing IVRA, 30 mL saline was simultaneously administered to the systemic circulation. All solutions were prepared by resident anesthesiologists, who were blinded to the study, using identical injectors.

The patients received premedication 45 min before the surgery with intramuscular 0.07 mg/kg midazolam and 0.01 mg/kg atropine. Two intravenous cannulas, one into the vein in the dorsal aspect of the hand that would undergo surgery and the other into the vein in the dorsal aspect of the opposite hand, were inserted for crystalloid infusion. The arm that would undergo surgery was elevated for 2 min and Esmarch's bandage was used to control blood flow. A double pneumatic tourniquet was placed around the upper arm and the proximal cuff was inflated to 250 mmHg. The absence of radial artery pulse in the arm isolated from the circulation was confirmed by the disappearance of pulse oximeter waves in the index finger of the same hand. The solutions, which were pre-prepared according to the groups defined above, were injected to the patients for over 90 s by an anesthesiologist blinded to the contents of drugs.

After the injection, the sensorial block was assessed every 30 s until the initiation of surgery by pinprick test using 22 gauge needle on the radial, ulnar and median nerve stimulation areas of the hand and of the anterior surface of the arm. Motor function was checked by asking the patient to bring the wrist and finger to extension and flexion and the time of complete motor block was recorded when spontaneous movement was impossible. The time elapsed from the injection of the study drug until the sensorial block was provided in all stimulation areas was recorded as the onset time of sensorial block. Likewise, the time elapsed from the injection of the study drug until achieving the complete motor block was recorded as the onset time of motor block. After achieving complete motor block and sensorial block, the distal tourniquet was inflated to 250 mmHg, the proximal tourniquet was deflated, and the surgical procedure was initiated. Mean arterial pressure (MAP), oxygen saturation (SpO2), and heart rate (HR) were monitored during the surgery, before and after tourniquet application, and until disappearance of anesthesia after deflating the tourniquet.

Pain level of the patients was assessed by 10 cm visual analogue scale (VAS; 0=no pain; 10=very severe pain). VAS scores were recorded before and after tourniquet application as well as at 5th, 10th, 15th, 20th, 30th, 40th, and 50th min during the surgery. If the patient had a VAS score of >4 and if required, 1 μg/kg fentanyl was administered for analgesia and the dosage and time were recorded.

The tourniquet was not deflated earlier than 30 min and it was not inflated more than 2 h. Tourniquet deflation after the surgery was performed by periodic deflation technique. The time of sensorial recovery was recorded (the time elapsed from the deflation of tourniquet to the highest pain felt by the patient via pinprick test performed every 30 s in all stimulation areas). The time of motor block recovery (time elapsed from the deflation of tourniquet to the spontaneous movement of the fingers) was also recorded.

The patients were monitored in the postoperative care unit for the first 2 h and then in the observation room for 24 h by anesthesiologists who were blinded to the study. MAP, HR, SpO2 monitoring and VAS measurement were performed at the postoperative 1st, 2nd, 4th, 6th, 12th, and 24th h. The patients with a VAS score of >4 were administered with 75 mg diclofenac sodium via intramuscular route. Analgesia requirement was recorded as duration and dosage.

The patients were monitored for intraoperative and postoperative complications. In the event of hypotension (systolic arterial pressure <90 mmHg or a decrease of more than 50 mmHg from the normal value) during the surgery, 5 mg intravenous ephedrine was administered. In case of bradycardia (HR <50/min), 0.5 mg intravenous atropine was administered. Intravenous 4 mg ondansetron was administered for nausea and vomiting and oxygen was supplied via a facial mask when SpO2 decreased by more than 91%.

An anesthesiologist and a surgeon, who were blinded to the content of study drug, assessed the quality of anesthesia at the end of surgery as follows: 4: excellent, patient does not complain; 3: good, patient complains a little, no need for supplemental analgesic; 2: moderate, patient complains, need for supplemental analgesic; 1: failed, need for general anesthesia.

The Predictive Analytics Software (PASW) version 18.0 for Windows program (SPSS Inc., Chicago, USA) was used for statistical analysis. Descriptive statistics were expressed as number and percentage for categorical variables and as mean, standard deviation, median, the 25th percentile (Q1: the first quartile), and the 75th percentile (Q3: the third quartile) for numerical variables. For numerical variables, independent multiple group comparisons were performed by Kruskal-Wallis test for non-normally distributed data and by t-test for normally distributed data. Mann-Whitney U test with Bonferroni correction was used for subgroup analysis of non-normally distributed numerical variables. For multiple group comparisons of categorical variables, Chi-square test statistics was used in case the assumption of chi-square test was met, whereas Fisher's Exact test was used in case the assumption of chi-square test was not met. A p value of <0.05 was considered statistically significant.

With the assumption that the difference in the VAS score at the 5th min between the two surgical techniques being 1 and the expected standard deviation for two groups being 0.9, it was estimated to include 20 patients in the groups for which the least difference was expected. The statistical significance level was calculated as 0.015 owing to the presence of 3 groups and with the prediction that repeated measurement analysis would be performed assuming that the Bonferroni correction would be used. The power of the present study was 80% with these calculations.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-II patients who were planned to undergo hand surgery.

Exclusion Criteria:

* Patients with Raynaud's disease, those with sickle-cell anemia, and those receiving any drug for history of allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Onset time of sensory block | The sensorial block was assessed from the injection of the study drug until the initiation of surgery by pinprick test (approximately 175 seconds)
  After the injection, the sensorial block was assessed until the initiation of surgery by pinprick test using 22 gauge needle on the radial, ulnar and median nerve stimulation areas of the hand and of the anterior surface of the arm. The time elapsed from the injection of the study drug until the sensorial block was provided in all stimulation areas was recorded as the onset time of sensorial block.
Recovery time of sensory block | The time elapsed from the deflation of tourniquet to the highest pain felt by the patient via pinprick test (approximately 135 seconds)
  The time of sensorial recovery was recorded (the time elapsed from the deflation of tourniquet to the highest pain felt by the patient via pinprick test in all stimulation areas).
Onset time of motor block | The time elapsed from the injection of the study drug until achieving the complete motor block was recorded as the onset time of motor block (approximately 220 seconds)
Recovery time of motor block | Time elapsed from the deflation of tourniquet to the spontaneous movement of the fingers (approximately 165 seconds)

SECONDARY OUTCOMES:
Degree of intraoperative pain | VAS scores were recorded before (one minute ago) and after tourniquet (five minutes later) application as well as at 5th, 10th, 15th, 20th, 30th, 40th, and 50th min during the surgery
  Pain level of the patients was assessed by 10 cm visual analogue scale (VAS; 0=no pain; 10=very severe pain) for once throughout the study.There is no follow up visit in the study. VAS scores were recorded before (one minute ago) and after tourniquet (five minutes later) application as well as at 5th, 10th, 15th, 20th, 30th, 40th, and 50th min during the surgery for once throughout the study.
Degree of postoperative pain with VAS measurement | VAS measurement was performed at the postoperative 1st, 2nd, 4th, 6th, 12th and 24th hour.
  The patients were monitored in the postoperative care unit for the first 2 h and then in the observation room for 24 h by anesthesiologists who were blinded to the study. VAS measurement was performed at the postoperative 1st, 2nd, 4th, 6th, 12th and 24th h for once throughout the study.There is no follow up visit in the study.
Quality of anesthesia | From the initiation of surgery (30 minutes) up to 24 hours after surgery, an average of 24,5 hours
  Quality of anesthesia is assessed as follows. 4: excellent, patient does not complain; 3: good, patient complains a little, no need for supplemental analgesic; 2: moderate, patient complains, need for supplemental analgesic; 1: failed, need for general anesthesia

REFERENCES:
- [Background] Chan VW, Peng PW, Kaszas Z, Middleton WJ, Muni R, Anastakis DG, Graham BA. A comparative study of general anesthesia, intravenous regional anesthesia, and axillary block for outpatient hand surgery: clinical outcome and cost analysis. Anesth Analg. 2001 Nov;93(5):1181-4. doi: 10.1097/00000539-200111000-00025. PMID 11682392
- [Background] dos Reis A Jr. Intravenous regional anesthesia--first century (1908-2008). Beggining, development, and current status. Rev Bras Anestesiol. 2008 May-Jun;58(3):299-321. doi: 10.1590/s0034-70942008000300013. English, Portuguese. PMID 19378526
- [Background] Choyce A, Peng P. A systematic review of adjuncts for intravenous regional anesthesia for surgical procedures. Can J Anaesth. 2002 Jan;49(1):32-45. doi: 10.1007/BF03020416. PMID 11782326
- [Background] Vazzana M, Andreani T, Fangueiro J, Faggio C, Silva C, Santini A, Garcia ML, Silva AM, Souto EB. Tramadol hydrochloride: pharmacokinetics, pharmacodynamics, adverse side effects, co-administration of drugs and new drug delivery systems. Biomed Pharmacother. 2015 Mar;70:234-8. doi: 10.1016/j.biopha.2015.01.022. Epub 2015 Feb 7. PMID 25776506
- [Background] Pang WW, Mok MS, Chang DP, Huang MH. Local anesthetic effect of tramadol, metoclopramide, and lidocaine following intradermal injection. Reg Anesth Pain Med. 1998 Nov-Dec;23(6):580-3. doi: 10.1016/s1098-7339(98)90085-2. PMID 9840854
- [Background] Pang WW, Huang PY, Chang DP, Huang MH. The peripheral analgesic effect of tramadol in reducing propofol injection pain: a comparison with lidocaine. Reg Anesth Pain Med. 1999 May-Jun;24(3):246-9. doi: 10.1016/s1098-7339(99)90136-0. PMID 10338176
- [Background] Sousa AM, Ashmawi HA, Costa LS, Posso IP, Slullitel A. Percutaneous sciatic nerve block with tramadol induces analgesia and motor blockade in two animal pain models. Braz J Med Biol Res. 2012 Feb;45(2):147-52. doi: 10.1590/s0100-879x2011007500164. Epub 2011 Dec 23. PMID 22183244
- [Background] Kapral S, Gollmann G, Waltl B, Likar R, Sladen RN, Weinstabl C, Lehofer F. Tramadol added to mepivacaine prolongs the duration of an axillary brachial plexus blockade. Anesth Analg. 1999 Apr;88(4):853-6. doi: 10.1097/00000539-199904000-00032. PMID 10195537
- [Background] Nagpal V, Rana S, Singh J, Chaudhary SK. Comparative study of systemically and perineurally administered tramadol as an adjunct for supraclavicular brachial plexus block. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):191-5. doi: 10.4103/0970-9185.155147. PMID 25948899
- [Background] Bigat Z, Boztug N, Hadimioglu N, Cete N, Coskunfirat N, Ertok E. Does dexamethasone improve the quality of intravenous regional anesthesia and analgesia? A randomized, controlled clinical study. Anesth Analg. 2006 Feb;102(2):605-9. doi: 10.1213/01.ane.0000194944.54073.dd. PMID 16428570
- [Background] Kashefi P, Montazeri K, Honarmand A, Safavi M, Hosseini HM. The analgesic effect of midazolam when added to lidocaine for intravenous regional anaesthesia. J Res Med Sci. 2011 Sep;16(9):1139-48. PMID 22973382
- [Background] Khanna P, Mohan VK, Sunder RA. Efficacy of diltiazem as an adjunct to lignocaine in intravenous regional anesthesia. Saudi J Anaesth. 2013 Jul;7(3):305-9. doi: 10.4103/1658-354X.115359. PMID 24015135
- [Background] Memis D, Turan A, Karamanlioglu B, Pamukcu Z, Kurt I. Adding dexmedetomidine to lidocaine for intravenous regional anesthesia. Anesth Analg. 2004 Mar;98(3):835-40, table of contents. doi: 10.1213/01.ane.0000100680.77978.66. PMID 14980948
- [Background] Sen H, Kulahci Y, Bicerer E, Ozkan S, Dagli G, Turan A. The analgesic effect of paracetamol when added to lidocaine for intravenous regional anesthesia. Anesth Analg. 2009 Oct;109(4):1327-30. doi: 10.1213/ane.0b013e3181b0fedb. PMID 19762765
- [Background] Sen S, Ugur B, Aydin ON, Ogurlu M, Gezer E, Savk O. The analgesic effect of lornoxicam when added to lidocaine for intravenous regional anaesthesia. Br J Anaesth. 2006 Sep;97(3):408-13. doi: 10.1093/bja/ael170. Epub 2006 Jul 15. PMID 16845131
- [Background] Sertoz N, Kocaoglu N, Ayanoglu HO. Comparison of lornoxicam and fentanyl when added to lidocaine in intravenous regional anesthesia. Braz J Anesthesiol. 2013 Jul-Aug;63(4):311-6. doi: 10.1016/j.bjane.2012.07.001. Epub 2013 Aug 13. PMID 24565236
- [Background] Sen S, Ugur B, Aydin ON, Ogurlu M, Gursoy F, Savk O. The analgesic effect of nitroglycerin added to lidocaine on intravenous regional anesthesia. Anesth Analg. 2006 Mar;102(3):916-20. doi: 10.1213/01.ane.0000195581.74190.48. PMID 16492852
- [Background] Turan A, Memis D, Karamanlioglu B, Guler T, Pamukcu Z. Intravenous regional anesthesia using lidocaine and magnesium. Anesth Analg. 2005 Apr;100(4):1189-1192. doi: 10.1213/01.ANE.0000145062.39112.C5. PMID 15781543
- [Background] Viscomi CM, Friend A, Parker C, Murphy T, Yarnell M. Ketamine as an adjuvant in lidocaine intravenous regional anesthesia: a randomized, double-blind, systemic control trial. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):130-3. doi: 10.1097/AAP.0b013e31819bb006. PMID 19282713
- [Background] Acalovschi I, Cristea T, Margarit S, Gavrus R. Tramadol added to lidocaine for intravenous regional anesthesia. Anesth Analg. 2001 Jan;92(1):209-14. doi: 10.1097/00000539-200101000-00040. PMID 11133629
- [Background] Aslan B, Izdes S, Kesimci E, Gumus T, Kanbak O. [Comparison of the effects of lidocaine, lidocaine plus tramadol and lidocaine plus morphine for intravenous regional anesthesia]. Agri. 2009 Jan;21(1):22-8. Turkish. PMID 19357997
- [Background] Alayurt S, Memis D, Pamukcu Z. The addition of sufentanil, tramadol or clonidine to lignocaine for intravenous regional anaesthesia. Anaesth Intensive Care. 2004 Feb;32(1):22-7. doi: 10.1177/0310057X0403200103. PMID 15058116
- [Background] Langlois G, Estebe JP, Gentili ME, Kerdiles L, Mouilleron P, Ecoffey C. The addition of tramadol to lidocaine does not reduce tourniquet and postoperative pain during iv regional anesthesia. Can J Anaesth. 2002 Feb;49(2):165-8. doi: 10.1007/BF03020489. PMID 11823394
- [Background] Tan SM, Pay LL, Chan ST. Intravenous regional anaesthesia using lignocaine and tramadol. Ann Acad Med Singap. 2001 Sep;30(5):516-9. PMID 11603137
- [Background] Siddiqui AK, Mowafi HA, Al-Ghamdi A, Ismail SA, AbuZeid HA. Tramadol as an adjuvant to intravenous regional anesthesia with lignocaine. Saudi Med J. 2008 Aug;29(8):1151-5. PMID 18690309
- [Background] Flamer D, Peng PW. Intravenous regional anesthesia: a review of common local anesthetic options and the use of opioids and muscle relaxants as adjuncts. Local Reg Anesth. 2011;4:57-76. doi: 10.2147/LRA.S16683. Epub 2011 Nov 25. PMID 22915894
- [Background] Grond S, Sablotzki A. Clinical pharmacology of tramadol. Clin Pharmacokinet. 2004;43(13):879-923. doi: 10.2165/00003088-200443130-00004. PMID 15509185